CLINICAL TRIAL: NCT04506164
Title: Effectiveness and Implementation of eScreening in Post 9/11 Transition Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SDR 19-443; 1I01HX003079-01A1 (NIH)
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Depression; Stress Disorders, Post-Traumatic; Suicide
Keywords: suicide; mental health; screening; technology; self report; veterans
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Suicide; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: his stepped-wedge trial relies on sequential roll-out to participating sites over time, while using other sites as controls until they begin implementation and facilitation. The eight participating sites will be stratified by size (a combination of number of TCM staff and average number of post-9/11 Veterans enrolled per month) and block randomized to four step/crossover cohorts of two sites each. All sites receive the same intervention at different times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stepped-wedge (Other): This stepped-wedge trial relies on sequential roll-out of eScreening to participating sites over time, while using other sites as controls until they begin implementation.
  Interventions: Other: Multicomponent Implementation Strategy; Other: eScreening

INTERVENTIONS:
Other: Multicomponent Implementation Strategy — The eScreening MCIS was developed over the past seven years and consists of: 1) eScreening software provision, 2) training, 3) RPIW, and 4) ongoing blended facilitation. The investigators developed our MCIS to address specific eScreening implementation barriers found in the investigators' prior research.
Other: eScreening — eScreening is a clinical patient self report system that allows Veterans to complete clinical reminders and other self report screens using a secure connection from any internet connected device.

SUMMARY:
Electronic screening is effective for timely detection of, and intervention for, suicidal ideation and other mental health symptoms. The VA eScreening program is a patient self-report electronic screening system that has shown promise for the efficient and effective collection of mental and physical health information among Veterans. However, additional effectiveness and implementation research is warranted to evaluate the impact of eScreening within VHA. This study will address questions of the impact of eScreening compared to screening as usual, while evaluating a multi-component implementation strategy (MCIS) for optimal enterprise rollout of eScreening in VA Transition Care Management clinics.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness and implementation of an electronic screening program called eScreening compared to standard of care paper and/or verbal screening methods in VHA Transition Care Management (TCM) programs. This is a mixed methods hybrid 2, effectiveness-implementation, stepped-wedge (SW) trial of eScreening in eight sites. The following eight sites are implementation sites where no research-related activities will be conducted: Oklahoma City VA Health Care System, Chillicothe VA Medical Center, Orlando VA Medical Center, VA Western Colorado Health Care System, VA Puget Sound Health Care System, Roseburg VA Health Care System, VA Salt Lake City Health Care System, West Palm Beach VA Medical Center. These sites will implement screening as part of routine clinical care. They will not collect data and will not obtain independent IRB approval.

Study investigators will collect the following data:

EMR data: EMR data will extracted from the Corporate Data Warehouse (CDW) database. EMR data will consist of 1) the number of Veterans that enrolled in the healthcare system and the date and time they enrolled (144 Veterans average per month across sites), 2) the date and time that they received PC-PTSD-5+I9, PHQ-2 +I9, AUDIT-C, CSSR-S, and the disposition (positive/negative screen), 3) date and time they received comprehensive suicide risk evaluation (CSRE), and 4) mental health care referrals. These data will be used to calculate the overall rate of screening completion and referral to mental health care and the average length of time to screening completion. The investigators will also collect age, sex, race, and ethnicity data to include as covariates in the models.

eScreening system: the investigators will use the eScreening reports functionality to pull eScreening usage data for the sites.

Staff participants: approximately 4-8 Transition Care Management staff (primarily social workers, but could include Medical Support Assistants or other professionals) at each of the 8 VHA sites who have direct or indirect involvement with implementation of eScreening will be asked to take part in this research. Participation will involve one 30-minute individual telephone survey/interview, two 60-minute individual telephone interviews, and one 20-minute online survey. The interviews and surveys will focus on assessing the feasibility and acceptability of the eScreening implementation strategy; factors affecting adoption, implementation, and sustained use of eScreening; and post implementation outcomes. All data from staff will be collected virtually.

The following is a detailed description of the study procedures, timeline, data, and analyses.

After a 6-month start up period involving planning and site randomization, the stepped-wedge trial will begin. This stepped-wedge trial relies on sequential roll-out to participating sites over time, while using other sites as controls until they begin implementation and facilitation. The eight participating sites will be stratified by size (a combination of number of TCM staff and average number of post-9/11 Veterans enrolled per month) and block randomized to four step/crossover cohorts of two sites each. All step/crossover cohorts will go through a 3-month pre-implementation (Pre-Imp) phase, followed by a 9-month active implementation using the eScreening MCIS. The eScreening MCIS will begin with a 3-month period that will include eScreening software provision, training, RPIW, and blended facilitation followed by 6 months of ongoing blended facilitation (9 months total). After the active implementation, all sites will have a 9-month sustainment period. Multiple types of data will be collected, including electronic medical record data, staff measures and interviews, field notes, and time motion tracking (described below). Data collection will begin at pre-implementation for each site and continue through sustainment.

Study Start up (0 to 6 months):

Randomization and internal facilitators. Sites will be stratified by size, block randomized into four step/crossover cohorts, and engaged in selecting the internal facilitators, who will be serving as site eScreening implementation champions during the study. During site selection, the investigators identified champions who support the use of eScreening and who have established relationships with the TCM team.

Finalize Materials. The qualitative lead co-investigator along with the PI and the implementation science expert will guide the development and pilot testing of the study questionnaires, time and adaptation trackers, and interview guides using PRISM.

Lean/Six Sigma RPIW training. The investigators' team has over 7 years of experience implementing eScreening in diverse clinical settings, using the RPIW approach. To prepare for formal RPIW facilitation, two external facilitators will be trained to facilitate eScreening RPIWs, including the primary facilitator (master's level) and a backup (the PI) by a blackbelt level Lean/Six Sigma expert in the Systems Redesign program at San Diego Healthcare System. As part of the training, the external facilitators will facilitate two formal eScreening RPIWs with implementation sites not participating in the study.

Finalize training materials. The investigators' team has developed an eScreening VA Pulse Site to make accessing technical information and training materials easy for staff. The site includes frequently asked questions, tutorial videos, a technical manual and user guide, a large amount of training information, and the eScreening playbook. In collaboration with the eScreening OIT team, the investigators will update these materials to include the most recent information on eScreening and to support the training protocol.

Stakeholder Meeting: Building upon several preliminary meetings with national and facility stakeholders, the investigators will host a formal teleconference start-up meeting with National TCM leadership, site internal facilitators, VA OIT eScreening Program Manager, VA Innovations staff, and the PI and co-investigators and research staff. The aim of this meeting is to orient everyone to the goals of the study, communicate the national stakeholder preferences for the content and frequency of interactions, and identify and address possible logistical barriers and facilitators. The 2-hour meeting will use a storyboard format to describe procedures and generate discussion through a structured focus group format employed in prior work. These meetings will occur every six months during the study. An external VHA advisory group, which includes Veterans, will review the research materials and plan.

Stepped-Wedge Trial (7 to 45 months):

Based on preliminary work, the investigators anticipate a sample of 45 TCM and related staff will be enrolled in this study. Patient level data will be collected from EMR (for which the investigators will apply for a HIPPA waiver), and no Veterans will directly participate. Recruitment procedures will be reviewed, and adjusted, if needed, in the startup period, but the proposed procedure will be as follows: 1) Internal facilitators, TCM staff and eScreening implementation-related stakeholder staff at each site will be invited to participate in the study; 2) An informational session about the study's leadership and purpose, selection of participants, and use of data will be conducted. Potential staff participants will be informed that their participation is entirely voluntary and their decision about participation will not affect their employment, merit, or promotion. Following this informational session, research staff consent interested participants. After consent has been signed, enrolled staff members will receive a link to an online survey and will be scheduled for a preliminary interview by the evaluation lead. If staff turnover occurs, the investigators will attempt to assess the staff member prior to leaving and replace and train another participant with similar functions within the clinic. Each of the four step/crossover cohorts will go through the following phases sequentially during the study.

Pre-implementation (Pre-Imp) phase. This phase will last 3 months during which the research team will work with the internal facilitators to: 1) gather pre-implementation information including detailed information on the processes in place for TCM screening upon enrollment ; 2) identify points of contact for iPads and other logistical needs; 3) establish communication with TCM staff and others working with the TCM staff; 4) recruit staff participants for the study; and 5) begin ongoing tracking of process data from field notes and time motion tracking. TCM staff names, clinic names, note titles, scheduling the RPIW, and clinical reminders completed by program staff will be gathered and used for subsequent development of user accounts and content customization during the implementation phase. The implementation team will also provide psychoeducation to the staff on the importance of screening. This phase will serve as an attention control condition to which the baseline control and intervention conditions will be compared.

During pre-implementation, TCM teams will continue usual screening procedures. These involve interview or self-report, paper-based collection of post-9/11 screening measures, including the system-wide standardized assessments of depression, PTSD and alcohol use (PHQ-2 +I9, PCPTSD +I9, and Audit-C, respectively). Patients who score positive on the PHQ-2 +I9, PCPTSD +I9 are then administered the Columbia Suicide Severity Rating Scale (C-SSRS), which collects more information regarding risk of suicide. Veterans who are positive on C-SSRS then receive a Comprehensive Suicide Risk Evaluation and are referred for appropriate follow-up. A detailed description and flow map of the current screening process at each site will be developed by the external facilitator (research team) and internal facilitator (site staff) with information from the TCM staff prior to the implementation phase.

Active Implementation (MCIS): The eScreening MCIS was developed over the past seven years and consists of: 1) eScreening software provision, 2) training, 3) RPIW, and 4) ongoing blended facilitation. The investigators developed the MCIS to address specific eScreening implementation barriers found in prior research. In order to address system level barriers related to OIT support, the investigators developed a technical support infrastructure for eScreening using existing VA IT resources (see LOS) as part of eScreening provision. The training component addresses educational barriers regarding eScreening use and the research available. Blended facilitation also addressed educational barriers as well as, technology related and other unforeseen challenges. The RPIW process will address, leadership support, staff buy-in, resources needed and by engaging all stakeholders in the process and developing a site-specific and clear plan for implementation. The RPIW specifically includes a section where the team generates possible barriers and solutions in day 2.

eScreening. eScreening is a VHA program that allows Veterans to answer self-report screening questions via an iPad connected to the VHA secure Wi-Fi. eScreening reads from and writes to the VHA EMR. The highlighted features of eScreening include: 1) the ability for Veterans to enter screening information directly without the involvement of a clinician; 2) immediate scoring of measures; 3) an editable note generated in the EMR; and 4) clinician alerts for positive mental health screens that require follow-up for suicide risk.

Training. eScreening training will be virtual and asynchronous and include a 1-hour instructional PowerPoint that will be presented by the external facilitator. The PowerPoint is followed by an hour of tutorial videos showing all steps of (creating assessments, adding Veterans, saving to VistA, searching for assessments, creating scheduled appointment assessments, accessing reports). Hands-on training for users will be available in group format or individually by the training staff as requested by the TCM site staff. Additional training materials can be accessed via the eScreening Pulse site which include a series of quick guides to address eScreening customization, assessment set-up and dashboard use. Frequently asked questions will also be available on the Pulse site.

RPIW. The 3-day RPIW will facilitated virtually by the external facilitator with assistance from the onsite internal facilitator and will include the TCM team, related staff (i.e., medical support staff, clerks), and other site stakeholders. The first day of the process will train participants in the RPIW principles and will introduce a summary of the information gathered in the Pre-Implementation Phase, including a graphic of the current state process map which will then be refined and finalized. The second day consists of collective efforts to map a targeted future state, conduct a gap analysis, and identifying relevant factors and barriers unique to the site. The third day is dedicated to the repetition of action planning, execution, and reevaluation to finalize the targeted state and identify clinically meaningful goals for improvement. Using a Plan-Do-Study-Act (PDSA) framework, the plans to achieve the target state are enacted with a detailed plan that includes who, what, when for each step in the plan. Due to the flexibility of eScreening and the implementation strategy, each TCM program may choose to integrate eScreening into their workflow based on the specific needs of their program, available resources, and other factors.

Blended facilitation. Blended facilitation will include a primary external facilitator from the eScreening team who will work with the site internal facilitator to schedule meetings, training sessions, and phone calls. The external facilitator will be the main point of contact for implementation-related questions. The internal facilitator, selected during the startup period, will work with the external facilitator to navigate internal site systems (i.e., local leadership, OIT, logistics) and serve as a champion for the eScreening project at each site.

Overview of Data Sources & Timing for Data Collection:

The study will use a mixed-methods design and will collect a combination of quantitative and qualitative data from multiple stakeholders and at multiple time points. A general overview of the data sources and data collection time points are provided in this section. More specific data collection and analysis considerations are provided under each aim.

Quantitative data sources and timing for data collection. Quantitative data collection includes data from the EMR, the eScreening system, and surveys that will be completed by staff participants. The investigators will extract EMR data at the beginning and end of Pre-Imp, at the end of the MCIS period, and at 9 months post-MCIS. The investigators will use the eScreening reports functionality to pull eScreening usage data for each cohort after the MCIS period and 9 months post-MCIS. The investigators will conduct a Pre-Imp individual telephone survey/interview using the feasibility and acceptability scales developed by Weiner et al (2017). The investigators will also use a secure online survey system (i.e., Qualtrics or RedCap) to collect survey elements based on the PRISM and its RE-AIM outcomes after the active implementation phase.

Qualitative data sources and timing for data collection. Qualitative data will be collected using field notes and interviews. The investigators will take field notes using a structured template during telephone meetings/calls throughout the pre-implementation and implementation stages including initial contact, during the RPIW, and the facilitation contact sessions. Research staff will take extensive field notes to describe the clinical environment, work flows, patient population, and relational atmosphere. Individual telephone interviews will be conducted with purposefully selected site staff during pre-implementation, post-implementation, and the sustainment phase. Interviews will focus on factors affecting adoption, implementation, and sustained use of eScreening. Both mindset and practical issues will be explored to illustrate implementation issues, challenges, and underpinnings of success. A specific set of probes will outline, and diagram tasks involved step-by-step to document barriers and facilitators and when communication and coordination were needed.

Aim 1 Data collection and analyses:

Aim 1: Evaluate eScreening, compared to paper and verbal screening, guided by the RE-AIM outcomes of PRISM in 8 TCM programs, using a cluster randomized, stepped wedge design. Hypothesis 1 (Reach): Compared to paper and verbal screening, eScreening will yield a significantly higher rate of screening. Hypothesis 2 (Effectiveness): 2a: Compared to paper and verbal screening, eScreening will result in significantly less time for mental health and suicide screening. 2b: Compared to paper and verbal screening, eScreening will result in significantly higher rate of referral to needed care.

Data collection. The investigators will obtain a HIPAA waiver to collect the following data: 1) the number of Veterans that enrolled in the healthcare system and the date and time they enrolled (144 Veterans average per month across sites), 2) the date and time that they received PC-PTSD-5+I9, PHQ-2 +I9, AUDIT-C, CSSR-S, and the disposition (positive/negative screen), 3) date and time they received comprehensive suicide risk evaluation (CSRE), and 4) mental health care referrals. These data will be used to calculate the overall rate of screening completion and referral to mental health care during the baseline control period and the average length of time to screening completion. The same data will be collected for the previous nine months post- implementation and sustainment. Based on the average enrollment data for the investigators' sites over the past year, approximately 27,600 Veterans will enroll in VA healthcare during the 27-month baseline control, Pre-Imp, post MCIS, and Sustainment data time-periods.

Sample size and power calculation: the investigators powered the study for the intervention effect of the effectiveness outcomes in Aim 1. The investigators assumed a common intervention effect across all cohorts/steps and Hierarchical Linear Modeling (HLM) to account for clustering, including a fixed effect for cohort/step of crossover to account for secular trends and an indicator of intervention phase change (e.g., control vs. intervention) to provide intervention effects. Power was calculated based on established methods for SW trials. The investigators set type I error rate alpha = 0.05, Cohen's d (or h for binary outcomes) effect size = 0.1, power = 0.8, and assumed an intraclass correlation (ICC) = 0.20, which is a conservative estimate based similar studies. Under these assumptions, the estimated sample size needed for the proposed study is approximately N = 5,000 participants. Data from the investigators' pilot study show effect sizes that are all above this detectable effect sizes. Given that 144 new post-9/11 Veterans are enrolled on average across implementation sites each month and the investigators will collect data at each site over a 24-month period, the study is sufficiently powered to detect effect sizes observed in similar studies.

Statistical analysis and hypothesis testing. Data analyses will proceed in stages and will follow the recommendations of the Prevention Science and Methodology Group for randomized field trials. Preliminary data screening and cleaning will require examination of the data distributions for normality and missing data patterns at both the univariate and multivariate level. Missing data are expected to be limited and are readily incorporated in HLM if the data can be assumed to be missing at random using Maximum Likelihood estimation. If the data are determined not to be missing at random, missing data mechanisms will be built into the target statistical models. HLM will be used as the primary statistical model due to the nested (or clustered) structure of the data (veterans [level 1] nested within TCM clinics [level 2] nested within implementation site [level 3]), with random assignment occurring at the implementation site level. HLM is a flexible modeling strategy that allows for the integration of fixed and random effects in nested/clustered data structures with normal and non-normal response variables. Demographic information about participants during the MCIS and control phases will be statistically compared within and between sites to ensure comparability. Any characteristics that differ between the intervention and control groups will be included as covariates in subsequent models to minimize bias. Fixed effects will be included in each model to account for study phase (i.e., baseline control, Pre-Imp/attention control, MCIS, and sustainment) and step/crossover cohort, to account for secular trends. The investigators will also be able to test interactions between study phase and step to determine whether intervention effects differed by cohort and whether intervention effects varied between TCM clinics within implementations sites. Separate models will be tested to determine whether a greater proportion of Veterans were screened for mental health and suicide risk (Reach) and referred to care (Effectiveness) during the MCIS and/or sustainment phases relative to the baseline and/or attention control phases. Additional models will test whether the mean number of days between enrollment and screening were lower (Effectiveness) during the MCIS and/or sustainment phases relative to the baseline and attention control phases. In all analyses, the investigators will set statistical significance at =0.05 and use Holm-Bonferroni adjustments for 5 tests and false discovery rate methods for >6 tests. When multiple correlated outcomes (dependent outcomes) are analyzed with each hypothesis, corrections will be calculated based on the effective number of independent tests when applying the multiple comparison procedures

Aim 2 Data collection and analyses:

Aim 2: Evaluate the feasibility, acceptability, and potential impact of the MCIS, guided by the RE-AIM outcomes of PRISM, adoption, implementation, and maintenance using mixed methods.

Data collection. The investigators will use a mixed methods approach and collect both quantitative and qualitative data guided by the RE-AIM outcomes of PRISM. For the replication cost, the investigators will use the a time tracker previously used for VA implementation efforts. The tool will be customized for this study and used to incrementally capture all facilitation activity by the external facilitator. Activities will then be quantified and used to develop a replication cost estimate by site.

Quantitative data analysis. The investigators will use descriptive statistics to summarize quantitative measures for each PRISM outcome using 50% as a benchmark. Adoption will be calculated as the overall number and proportion of TCM clinics that are willing to initiate eScreening, relative to the total number of TCM clinics across implementation sites and within each implementation site, as well as the overall number and proportion of providers who are willing to adopt eScreening relative to the total number of providers across implementation sites, across TCM clinics at each implementation site, and within each TCM clinic. Implementation will be calculated as the proportion of TCM clinics and providers within clinics who implement eScreening. The investigators will also calculate mean ratings of the acceptability and feasibility of the MCIS across providers within TCM clinics and across implementation sites. Time tracker data will be analyzed using the VA general ledger, which includes all labor costs including employee benefits and employer contributions to taxes. Indirect costs should be incurred in proportion to direct costs and will be estimated based on VA Health Economics Resource Center (HERC) guidance. Maintenance will be calculated as the proportion of TCM clinics and providers within clinics who implement eScreening during the sustainment phase (i.e., the 9-month period following initial implementation).

Qualitative data analysis. Study investigators or an experienced, trained member of the study team will conduct semi-structured interviews. Interviews will be audio recorded, transcribed by the VA CTSP, and entered into the qualitative software program, ATLAS.ti. A key aspect to this analysis is to answer these questions: What influences adoption of eScreening by providers? What factors influenced the implementation of eScreening? What factors promote maintenance? The analysis will also answer the bigger question of why providers do or do not implement eScreening, including understanding any practical clinic work flow reasons for use or non-use, or key underlying characteristics of eScreening program or provider. The analysis will consider emergent themes using an editing approach. Two project team members will independently code the semi-structured interview data collected. A third team member will assess coding quality and resolve conflicts.

Convergent analysis. Using a mixed-methods convergent design, the qualitative research core team will analyze the data concurrently with the quantitative data to explain and support/refute the quantitative data and add to insights regarding future implementation research and dissemination efforts.

Aim 3 Data collection and analyses:

Aim 3: Describe and compare high and low eScreening reach sites guided by contextual constructs of PRISM using qualitative comparative analysis to explore factors influencing the reach of eScreening and the use of the eScreening MCIS. In Aim 3, qualitative data from contextual elements of PRISM will be used to construct comparative analysis between high and low eScreening reach sites. Questions and measures assessing the PRISM contextual dimensions will be included in the proposed interviews and field notes (qualitative data) and will also be informed by the proposed surveys and EMR data (quantitative data).

Data analysis. Qualitative data will be analyzed as described for aim 2, but the investigators will use a template approach for the analysis using constructs from contextual factors. The investigators will use codes identified and created based on the PRISM constructs and other emergent themes to tag the relevant transcript quotations. Quotation reports will list the associated quotations verbatim by site. Sites will be divided by high vs. low reach using a cutoff score of 30% (from Aim 1), based on prior work. Qualitative comparative analysis (QCA) will allow us compare high and low eScreening reach sites to identify factors influencing the implementation of eScreening and the impact of the MCIS using systematic cross-case comparison to better understand causal complexity. The investigators will list and count different combinations of variables in the data set, and then apply logical inference rules to evaluate whether alternative inferences are supported by the data. Using the investigators' outcome of interest (i.e. high reach) and a list of conditions (i.e. contextual factors) that may be associated with that outcome the investigators will develop calibration metrics using a crisp dichotomous set. Calibration involves considering how each site is related to the pre-defined PRISM concept using specific decision rules. The investigators will establish a codebook detailing the conditions and decision rules. Third, the investigators will calibrate the data. Specifically, using coded data, each site will be calibrated dichotomously as either "having" (1.0) or "not having" (0.0) each condition. After the investigators' sites are calibrated, the investigators will construct a truth table, using Stata, to analyze logical combinations of conditions to determine if specific combinations share the outcome. Using Boolean logic, the investigators will minimize the truth table to arrive at pathways to the outcome. The pathways will then be assessed using the consistency and coverage parameters of fit. A thematic analysis of site interview data will be used to supplement QCA findings.

ELIGIBILITY:
Inclusion Criteria:

Staff inclusion criteria:

* Direct or indirect involvement with implementation of eScreening at the site
* Capable of informed consent

Exclusion Criteria:

Staff exclusion criteria:

* Not involved in or directly impacted by eScreening involvement at each site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in rate of screening completion | baseline (6-18months), post (18-27months), and followup (27-36months).
  Rate of screening completion will be calculated using medical record data from Veterans who enroll for care during the 3 months prior to the above time points. Rate of completed PC-PTSD-5+I9, PHQ-2 +I9, AUDIT-C, CSSR-S, and the disposition (positive/negative screen), 3) Rate of comprehensive suicide risk evaluation (CSRE) will be used. Change in rates between screening as usual (baseline) and eScreening will be evaluated over the timepoints.
Change in time to screening completion | baseline (6-18months), post (18-27months), and followup (27-36months).
  Time to screening completion will be calculated using medical record data from Veterans who enroll for care during the 3 months prior to the above time points. Date and time of enrollment date and time of PC-PTSD-5+I9, PHQ-2 +I9, AUDIT-C, CSSR-S, and the disposition (positive/negative screen), 3) date and time they received comprehensive suicide risk evaluation (CSRE) will be used. Speed will be calculated using time from enrollment to screening (minutes, hours, days). Change in speed between screening as usual (baseline) and eScreening will be evaluated over the timepoints.

SECONDARY OUTCOMES:
Change in rate of referral to care | baseline (6-18months), post (18-27months), and followup (27-36months).
  Rate of referral to follow up care will be collected from using medical record data from Veterans who enroll for care during the 3 months prior to the above time points. The percent of Veterans who enrolled and screen positive on the PC-PTSD-5+I9, PHQ-2 +I9, AUDIT-C, CSSR-S and are referred to additional care will be calculated. Change in rates between screening as usual (baseline) and eScreening will be evaluated over the timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: James Pittman, PhD MSW, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Only data sets without individual identifiers will be generated and shared.

REFERENCES:
- [Result] Pittman JOE, Lindamer L, Afari N, Depp C, Villodas M, Hamilton A, Kim B, Mor MK, Almklov E, Gault J, Rabin B. Implementing eScreening for suicide prevention in VA post-9/11 transition programs using a stepped-wedge, mixed-method, hybrid type-II implementation trial: a study protocol. Implement Sci Commun. 2021 Apr 29;2(1):46. doi: 10.1186/s43058-021-00142-9. PMID 33926577

DOCUMENTS (1):
  • Informed Consent Form (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT04506164/ICF_001.pdf